CLINICAL TRIAL: NCT03565991
Title: A PHASE 2 STUDY TO EVALUATE SAFETY AND ANTI-TUMOR ACTIVITY OF AVELUMAB IN COMBINATION WITH TALAZOPARIB IN PATIENTS WITH BRCA OR ATM MUTANT TUMORS JAVELIN BRCA/ATM
Brief Title: Javelin BRCA/ATM: Avelumab Plus Talazoparib in Patients With BRCA or ATM Mutant Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated since there was no need for further safety or efficacy data to be collected. The participants having benefit from the investigational treatments have been moved to a continuation study (NCT05059522)
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B9991032; 2018-000345-39 (EudraCT Number)
Record Dates: First submitted 2018-05-25; First posted 2018-06-21 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced or Metastatic Solid Tumors; Genes, BRCA 1
Keywords: BRCA, ATM
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — avelumab; talazoparib

STUDY DESIGN:
Intervention Model Description: Single arm study with two cohorts enrolled in parallel.
  * Cohort 1 will enroll patients with locally advanced or metastatic solid tumors with one or more defects in the BRCA1 or BRCA2 genes
  * Cohort 2 will enroll patients with locally advanced or metastatic solid tumors with one or more defects in the ATM gene
Masking Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination of avelumab and talazoparib (Experimental): Single arm open label
  Interventions: Drug: Avelumab; Drug: Talazoparib

INTERVENTIONS:
Drug: Avelumab — IV treatment
  Other Names: Bavencio
Drug: Talazoparib — Oral treatment
  Other Names: MDV3800, BMN 673

SUMMARY:
Avelumab in combination with talazoparib will be investigated in patients with locally advanced or metastatic solid tumors with a BRCA or ATM defect.

DETAILED DESCRIPTION:
Avelumab is a human immunoglobulin (Ig)G1 monoclonal antibody (mAb) directed against programmed death ligand 1 (PD-L1). Avelumab selectively binds to PD-L1 and competitively blocks its interaction with programmed death receptor 1 (PD-1), thereby interfering with this key immune checkpoint inhibition pathway. Avelumab is currently being investigated as single agent and in combination with other anti cancer therapies in patients with locally advanced or metastatic solid tumors and various hematological malignancies.

Talazoparib is a potent, orally bioavailable poly (adenosine diphosphate [ADP] ribose) polymerase (PARP) inhibitor, which is cytotoxic to human cancer cell lines harboring gene mutations that compromise deoxyribonucleic acid (DNA) repair, an effect referred to as synthetic lethality, and by trapping PARP protein on DNA thereby preventing DNA repair, replication, and transcription.

Avelumab in combination with talazoparib will be investigated in patients with locally advanced (primary or recurrent) or metastatic solid tumors with a BReast CAncer susceptibility gene (BRCA)1, or BRCA2, or ataxia telangiectasia mutated (ATM) gene defect.

ELIGIBILITY:
Inclusion Criteria:

* BRCA1, BRCA2 and/or ATM gene defect.
* Histological diagnosis of locally advanced (primary or recurrent) or metastatic solid tumors that are not amenable for treatment with curative intent
* Availability a tumor tissue sample from a diagnostic biopsy/surgery or a metastatic tumor biopsy.
* Progressive disease at study enrollment.
* Minimum age 18 years (in Japan, minimum age 20 years).
* ECOG performance status 0 or 1.
* Adequate bone marrow, renal and liver function.
* For childbearing female patients, negative serum or urine pregnancy test at screening
* Signed and dated informed consent document.

Exclusion Criteria:

* Prior anti-cancer therapy or radiation therapy within 2 weeks prior to enrolment. Palliative radiotherapy to metastatic lesion(s) permitted providing that it has been completed at least 2 days prior to enrolment and no significant toxicity are expected.
* Major surgery within 4 weeks prior to study enrollment.
* Current use of immunosuppressive medication at the time of study enrollment.
* Known prior severe hypersensitivity to investigational products or any component in their formulations
* Known history of immune-mediated colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis.
* Active or prior autoimmune disease that might deteriorate when receiving an immunostimulatory agent.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Administration of live attenuated vaccines within 4 weeks of study enrollment.
* Diagnosis of myelodysplastic syndrome.
* Known symptomatic brain metastases requiring steroids.
* Persisting toxicity related to prior therapy Grade >1.
* Known history of HIV or AIDS.
* Positive HBV or HCV test indicating acute or chronic infection.
* Active infection requiring systemic therapy.
* Clinically significant (active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months prior to study enrollment; unstable angina, congestive heart failure or a serious cardiac arrhythmia requiring medication.
* Diagnosis of any other malignancy within 2 years prior to study enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast, bladder, or cervix, or low-grade prostate cancer or other early-stage low-risk cancers.
* Pregnant or breastfeeding female patients; female or male patients who are able to have children who are unable or unwilling to use contraception as outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (97):
- United States (69):
  - Stanford Cancer Center, Palo Alto, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - Stanford Healthcare, Stanford, California
  - Stanford University School of Medicine, Stanford, California
  - Atlanta Cancer Care -Alpharetta, Alpharetta, Georgia
  - Northside Hospital, Inc. - GCS/Athens, Athens, Georgia
  - Northside Hospital, Inc. - GCS/Annex, Atlanta, Georgia
  - Atlanta Cancer Care - Atlanta, Atlanta, Georgia
  - Northside Hospital, Inc. - Central Research Department, Atlanta, Georgia
  - Northside Hospital, Inc. - GCS/Northside, Atlanta, Georgia
  - Northside Hospital, Inc. - GCS/Canton, Canton, Georgia
  - Atlanta Cancer Care - Cumming, Cumming, Georgia
  - Atlanta Cancer Care - Decatur, Decatur, Georgia
  - Northside Hospital, Inc.-GCS/Stemmer, Decatur, Georgia
  - Atlanta Cancer Care - Stockbridge, Jonesboro, Georgia
  - Northside Hospital, Inc.-GCS/Macon, Macon, Georgia
  - Northside Hospital, Inc.-GCS/Kennestone, Marietta, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer institute, Boston, Massachusetts
  - Siteman Cancer Center - St.Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Siteman Cancer Center - North County, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center- Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center- Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center - Investigational Drug Service Pharmacy, Long Island City, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - NY Investigational Pharmacy, New York, New York
  - NYU Langone Medical Center, New York, New York
  - NYU Langone Radiology - 32nd Street, New York, New York
  - NYU Langone Radiology Ambulatory Care Center East 41st Street, New York, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Rockefeller Outpatient Center, New York, New York
  - Rockefeller Outpatient Pavilion (53rd Street), New York, New York
  - Evelyn H. Lauder Breast and Imaging Center, New York, New York
  - Memorial Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - White Plains Hospital, White Plains, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Stephanie Spielman Comprehensive Breast Cancer, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio
  - OSU Gynecologic Oncology at Mill Run, Hilliard, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania/Penn Investigational Drug Services, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn IDS Central, Philadelphia, Pennsylvania
  - Magee-Women's Hospital Women's Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center Investigational Drug Service, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - The Sarah Cannon Research Institute, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Cleveland, Tennessee
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - The University of Texas, Houston, Texas
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense C
- France (3):
  - Centre Jean Perrin, Clermont-Ferrand
  - Groupe Hospitalier La Rochelle-Ré-Aunis, La Rochelle
  - Institut Regional du Cancer de Montpellier - ICM Val d'Aurelle, Montpellier
- Italy (8):
  - Presidio AO-U, Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi, Torette Di Ancona, AN
  - IRCCS-Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC
  - Azienda Socio-Sanitaria Territoriale Monza, Ospedale San Gerardo, Monza, MB
  - Fondazione IRCCS, Istituto Nazionale dei Tumori, Milan, MI
  - Istituto Europeo di Oncologia, Istituto di Ricovero e Cura a Carattere Scientifico, Milan, MI
  - Fondazione Pascale, IRCCS, Istituto Nazionale dei Tumori, Napoli
  - Azienda Policlinico Umberto I, Universita La Sapienza, Oncologia B, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Unità di Farmacologia Clinica, Roma
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Osaka International Cancer Institute, Osaka, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Netherlands (2):
  - Amsterdam University Medical Centre, location VUmc, Amsterdam, North Holland
  - Erasmus Universitair Medisch Centrum, Rotterdam, South Holland
- Spain (5):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - H.G.U. Gregorio Maranon, Madrid
  - Clinica Universidad de Navarra, Madrid
  - H.U. Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Virgen de Valme, Seville
- United Kingdom (2):
  - Barts Health NHS Trust, St Bartholomew's Hospital, London
  - Sarah Cannon Research Institute UK, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Schram AM, Colombo N, Arrowsmith E, Narayan V, Yonemori K, Scambia G, Zelnak A, Bauer TM, Jin N, Ulahannan SV, Colleoni M, Aftimos P, Donoghue MTA, Rosen E, Rudneva VA, Telli ML, Domchek SM, Galsky MD, Hoyle M, Chappey C, Stewart R, Blake-Haskins JA, Yap TA. Avelumab Plus Talazoparib in Patients With BRCA1/2- or ATM-Altered Advanced Solid Tumors: Results From JAVELIN BRCA/ATM, an Open-Label, Multicenter, Phase 2b, Tumor-Agnostic Trial. JAMA Oncol. 2023 Jan 1;9(1):29-39. doi: 10.1001/jamaoncol.2022.5218. PMID 36394867
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991032

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 270 participants were screened for this study, 202 participants were enrolled and assigned to study treatment but 2 participants never started the treatment. In total 200 participants were treated (159 in Cohort 1 and 41 in Cohort 2).
Groups:
- Cohort 1 (BReast CAncer Gene [BRCA] 1/2 Defect): Participants with locally advanced or metastatic solid tumors with one or more defects in the BRCA1 or BRCA2 genes were enrolled in Cohort 1. Talazoparib was self-administered orally at a starting dose of 1 mg Once Daily (QD) for participants with normal renal function or mild renal impairment until End of Treatment. Participants with moderate renal impairment received starting dose of 0.75 mg QD. Avelumab was administered as a 1-hour Intravenous (IV) infusion Every 2 Weeks (Q2W) on Days 1 and 15 of each 28-day cycle at a dose of 800 mg after administration of talazoparib and the premedication.
- Cohort 2 (Ataxia Telangiectasia Mutated [ATM] Defect): Participants with locally advanced or metastatic solid tumors with one or more defects in the ATM gene without concurrent BRCA1/2 defect were enrolled in Cohort 2. Talazoparib was self-administered orally at a starting dose of 1 mg QD for participants with normal renal function or mild renal impairment until End of Treatment. Participants with moderate renal impairment received starting dose of 0.75 mg QD. Avelumab was administered as a 1-hour IV infusion Q2W on Days 1 and 15 of each 28-day cycle at a dose of 800 mg after administration of talazoparib and the premedication.
Period: Overall Study
Arm/Group | Cohort 1 (BReast CAncer Gene [BRCA] 1/2 Defect) | Cohort 2 (Ataxia Telangiectasia Mutated [ATM] Defect)
Started | 159 | 41
Completed | 1 | 0
Not Completed | 158 | 41
Not completed — Other | 11 | 0
Not completed — Global deterioration of health status | 14 | 4
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Progressive disease | 121 | 29
Not completed — Death | 3 | 0
Not completed — Adverse Event | 7 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants who received at least 1 dose of study treatment.
Groups:
- Cohort 1 (BRCA 1/2 Defect): Participants with locally advanced or metastatic solid tumors with one or more defects in the BRCA1 or BRCA2 genes were enrolled in Cohort 1. Talazoparib was self-administered orally at a starting dose of 1 mg QD for participants with normal renal function or mild renal impairment until End of Treatment. Participants with moderate renal impairment received starting dose of 0.75 mg QD. Avelumab was administered as a 1-hour IV infusion Q2W on Days 1 and 15 of each 28-day cycle at a dose of 800 mg after administration of talazoparib and the premedication.
- Cohort 2 (ATM Defect): Participants with locally advanced or metastatic solid tumors with one or more defects in the ATM gene without concurrent BRCA1/2 defect were enrolled in Cohort 2. Talazoparib was self-administered orally at a starting dose of 1 mg QD for participants with normal renal function or mild renal impairment until End of Treatment. Participants with moderate renal impairment received starting dose of 0.75 mg QD. Avelumab was administered as a 1-hour IV infusion Q2W on Days 1 and 15 of each 28-day cycle at a dose of 800 mg after administration of talazoparib and the premedication.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect) | Total
Number analyzed (Participants) | 159 | 41 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.35 (12.88) | 61.76 (12.47) | 58.25 (12.89)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 110 | 25 | 135
  65 - <75 years | 34 | 11 | 45
  75 - <85 years | 15 | 3 | 18
  >=85 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 24 | 132
  Male | 51 | 17 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 2 | 13
  Not Hispanic or Latino | 131 | 39 | 170
  Unknown or Not Reported | 17 | 0 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 8 | 3 | 11
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 15 | 0 | 15
  White | 117 | 37 | 154
  Not reported | 18 | 1 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Objective Response (OR) as Assessed by Blinded Independent Central Review (BICR)
Description: For participants with solid tumors, except metastatic Castration Resistant Prostate Cancer (mCRPC), OR was defined as a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1), both confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. For participants with mCRPC, OR was defined as the percentage of participants with a best overall soft tissue response of CR or PR per RECIST v1.1 with no evidence of confirmed bone disease progression per Prostate Cancer Working Group 3 (PCWG3) criteria. Per RECIST v1.1, CR was defined as complete disappearance of all target and non-target lesions with the exception of nodal disease. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. Non-target PR lesions must be non-Progressive Disease (PD), where PD was unequivocal progression of pre-existing lesions.
Time Frame: From the first dose of study treatment until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to approximately 24 months
Population: The analysis set included all enrolled participants who received at least 1 dose of study treatment. Participants were classified according to the cohort assigned at enrollment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Percentage of participants | 27.7 [20.9 to 35.3] | 7.3 [1.5 to 19.9]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation where participants administered a product or medical device. TEAEs were those events with onset dates occurring during the on-treatment period. A Serious Adverse Event (SAE) was any untoward medical occurrence at any dose that: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or resulted in congenital anomaly/birth defect. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. TEAEs were graded by the investigator using National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) v4.03 as Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE.
Time Frame: From baseline up to 30 days after last dose of study treatment, maximum up to 4.3 years approximately
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Participants
  TEAEs | 156 | 40
  treatment-related TEAEs | 148 | 34
  grade >=3 TEAEs | 114 | 22
  grade >=3 treatment-related TEAEs | 85 | 17
  SAEs | 50 | 7
  treatment-related SAEs | 12 | 4
  TEAEs leading to discontinuation of all study drugs | 5 | 2
  treatment-related TEAEs leading to discontinuation of all study drugs | 0 | 1
  TEAEs leading to death | 14 | 2
  treatment-related TEAEs leading to death | 0 | 0

3. Secondary Outcome: Number of Participants With New or Worsening Hematology Laboratory Test Results During the On-Treatment Period
Description: The laboratory results were graded according to the CTCAE v4.03 severity grade whenever applicable. Laboratory test abnormalities were summarized according to worst toxicity grade observed for each laboratory test. As per NCI CTCAE toxicity grading v4.03, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE. On-treatment period was defined as the time from the first dose of study treatment through minimum (30 days + last dose of study treatment, start day of new anti-cancer drug therapy - 1 day).
Time Frame: From baseline up to 30 days after last dose of study treatment, maximum up to 4.3 years approximately
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study treatment. The number analyzed for each parameter in each treatment group was the number of participants evaluable for each parameter. Number of participants analyzed = participants evaluable for this outcome measure (OM), number analyzed = participants evaluable for the specific lab parameter per CTCAE criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Participants
  New or worsened to grade 1 (Parameter: activated partial thromboplastin time prolonged): number analyzed (Participants) | 5 | 1
  New or worsened to grade 1 (Parameter: activated partial thromboplastin time prolonged) | 0 | 0
  New or worsened to grade 2 (Parameter: activated partial thromboplastin time prolonged): number analyzed (Participants) | 5 | 1
  New or worsened to grade 2 (Parameter: activated partial thromboplastin time prolonged) | 0 | 0
  New or worsened to grade 3 (Parameter: activated partial thromboplastin time prolonged): number analyzed (Participants) | 5 | 1
  New or worsened to grade 3 (Parameter: activated partial thromboplastin time prolonged) | 0 | 0
  New or worsened to grade 4 (Parameter: activated partial thromboplastin time prolonged): number analyzed (Participants) | 5 | 1
  New or worsened to grade 4 (Parameter: activated partial thromboplastin time prolonged) | 0 | 0
  New or worsened to grade 1 (Parameter: anemia): number analyzed (Participants) | 151 | 40
  New or worsened to grade 1 (Parameter: anemia) | 27 | 9
  New or worsened to grade 2 (Parameter: anemia): number analyzed (Participants) | 151 | 40
  New or worsened to grade 2 (Parameter: anemia) | 33 | 6
  New or worsened to grade 3 (Parameter: anemia): number analyzed (Participants) | 151 | 40
  New or worsened to grade 3 (Parameter: anemia) | 61 | 12
  New or worsened to grade 4 (Parameter: anemia): number analyzed (Participants) | 151 | 40
  New or worsened to grade 4 (Parameter: anemia) | 0 | 0
  New or worsened to grade 1 (Parameter: hemoglobin increased): number analyzed (Participants) | 157 | 41
  New or worsened to grade 1 (Parameter: hemoglobin increased) | 1 | 0
  New or worsened to grade 2 (Parameter: hemoglobin increased): number analyzed (Participants) | 157 | 41
  New or worsened to grade 2 (Parameter: hemoglobin increased) | 0 | 0
  New or worsened to grade 3 (Parameter: hemoglobin increased): number analyzed (Participants) | 157 | 41
  New or worsened to grade 3 (Parameter: hemoglobin increased) | 0 | 0
  New or worsened to grade 4 (Parameter: hemoglobin increased): number analyzed (Participants) | 157 | 41
  New or worsened to grade 4 (Parameter: hemoglobin increased) | 0 | 0
  New or worsened to grade 1 (Parameter: International Normalized Ratio [INR] increased): number analyzed (Participants) | 6 | 0
  New or worsened to grade 1 (Parameter: International Normalized Ratio [INR] increased) | 1 | 0
  New or worsened to grade 2 (Parameter: INR increased): number analyzed (Participants) | 6 | 0
  New or worsened to grade 2 (Parameter: INR increased) | 0 | 0
  New or worsened to grade 3 (Parameter: INR increased): number analyzed (Participants) | 6 | 0
  New or worsened to grade 3 (Parameter: INR increased) | 0 | 0
  New or worsened to grade 4 (Parameter: INR increased): number analyzed (Participants) | 6 | 0
  New or worsened to grade 4 (Parameter: INR increased) | 0 | 0
  New or worsened to grade 1 (Parameter: lymphocyte count decreased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 1 (Parameter: lymphocyte count decreased) | 15 | 6
  New or worsened to grade 2 (Parameter: lymphocyte count decreased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 2 (Parameter: lymphocyte count decreased) | 58 | 15
  New or worsened to grade 3 (Parameter: lymphocyte count decreased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 3 (Parameter: lymphocyte count decreased) | 34 | 7
  New or worsened to grade 4 (Parameter: lymphocyte count decreased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 4 (Parameter: lymphocyte count decreased) | 3 | 0
  New or worsened to grade 1 (Parameter: lymphocyte count increased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 1 (Parameter: lymphocyte count increased) | 0 | 0
  New or worsened to grade 2 (Parameter: lymphocyte count increased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 2 (Parameter: lymphocyte count increased) | 3 | 0
  New or worsened to grade 3 (Parameter: lymphocyte count increased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 3 (Parameter: lymphocyte count increased) | 1 | 0
  New or worsened to grade 4 (Parameter: lymphocyte count increased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 4 (Parameter: lymphocyte count increased) | 0 | 0
  New or worsened to grade 1 (Parameter: neutrophil count decreased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 1 (Parameter: neutrophil count decreased) | 15 | 2
  New or worsened to grade 2 (Parameter: neutrophil count decreased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 2 (Parameter: neutrophil count decreased) | 42 | 8
  New or worsened to grade 3 (Parameter: neutrophil count decreased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 3 (Parameter: neutrophil count decreased) | 16 | 4
  New or worsened to grade 4 (Parameter: neutrophil count decreased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 4 (Parameter: neutrophil count decreased) | 3 | 1
  New or worsened to grade 1 (Parameter: platelet count decreased): number analyzed (Participants) | 152 | 41
  New or worsened to grade 1 (Parameter: platelet count decreased) | 59 | 16
  New or worsened to grade 2 (Parameter: platelet count decreased): number analyzed (Participants) | 152 | 41
  New or worsened to grade 2 (Parameter: platelet count decreased) | 16 | 3
  New or worsened to grade 3 (Parameter: platelet count decreased): number analyzed (Participants) | 152 | 41
  New or worsened to grade 3 (Parameter: platelet count decreased) | 14 | 4
  New or worsened to grade 4 (Parameter: platelet count decreased): number analyzed (Participants) | 152 | 41
  New or worsened to grade 4 (Parameter: platelet count decreased) | 11 | 1
  New or worsened to grade 1 (Parameter: white blood cell decreased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 1 (Parameter: white blood cell decreased) | 45 | 14
  New or worsened to grade 2 (Parameter: white blood cell decreased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 2 (Parameter: white blood cell decreased) | 52 | 11
  New or worsened to grade 3 (Parameter: white blood cell decreased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 3 (Parameter: white blood cell decreased) | 15 | 5
  New or worsened to grade 4 (Parameter: white blood cell decreased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 4 (Parameter: white blood cell decreased) | 2 | 0

4. Secondary Outcome: Number of Participants With New or Worsening Chemistry Laboratory Test Results During the On-Treatment Period
Description: as for outcome 3
Time Frame: From baseline up to 30 days after last dose of study treatment, maximum up to 4.3 years approximately
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Participants
  New or worsened to grade 1 (Parameter: alanine aminotransferase increased): number analyzed (Participants) | 152 | 41
  New or worsened to grade 1 (Parameter: alanine aminotransferase increased) | 30 | 10
  New or worsened to grade 2 (Parameter: alanine aminotransferase increased): number analyzed (Participants) | 152 | 41
  New or worsened to grade 2 (Parameter: alanine aminotransferase increased) | 6 | 0
  New or worsened to grade 3 (Parameter: alanine aminotransferase increased): number analyzed (Participants) | 152 | 41
  New or worsened to grade 3 (Parameter: alanine aminotransferase increased) | 3 | 3
  New or worsened to grade 4 (Parameter: alanine aminotransferase increased): number analyzed (Participants) | 152 | 41
  New or worsened to grade 4 (Parameter: alanine aminotransferase increased) | 1 | 0
  New or worsened to grade 1 (Parameter: alkaline phosphatase increased): number analyzed (Participants) | 153 | 41
  New or worsened to grade 1 (Parameter: alkaline phosphatase increased) | 25 | 12
  New or worsened to grade 2 (Parameter: alkaline phosphatase increased): number analyzed (Participants) | 153 | 41
  New or worsened to grade 2 (Parameter: alkaline phosphatase increased) | 21 | 5
  New or worsened to grade 3 (Parameter: alkaline phosphatase increased): number analyzed (Participants) | 153 | 41
  New or worsened to grade 3 (Parameter: alkaline phosphatase increased) | 7 | 1
  New or worsened to grade 4 (Parameter: alkaline phosphatase increased): number analyzed (Participants) | 153 | 41
  New or worsened to grade 4 (Parameter: alkaline phosphatase increased) | 1 | 0
  New or worsened to grade 1 (Parameter: aspartate aminotransferase increased): number analyzed (Participants) | 150 | 40
  New or worsened to grade 1 (Parameter: aspartate aminotransferase increased) | 35 | 5
  New or worsened to grade 2 (Parameter: aspartate aminotransferase increased): number analyzed (Participants) | 150 | 40
  New or worsened to grade 2 (Parameter: aspartate aminotransferase increased) | 13 | 2
  New or worsened to grade 3 (Parameter: aspartate aminotransferase increased): number analyzed (Participants) | 150 | 40
  New or worsened to grade 3 (Parameter: aspartate aminotransferase increased) | 2 | 4
  New or worsened to grade 4 (Parameter: aspartate aminotransferase increased): number analyzed (Participants) | 150 | 40
  New or worsened to grade 4 (Parameter: aspartate aminotransferase increased) | 1 | 0
  New or worsened to grade 1 (Parameter: blood bilirubin increased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 1 (Parameter: blood bilirubin increased) | 7 | 2
  New or worsened to grade 2 (Parameter: blood bilirubin increased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 2 (Parameter: blood bilirubin increased) | 7 | 2
  New or worsened to grade 3 (Parameter: blood bilirubin increased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 3 (Parameter: blood bilirubin increased) | 2 | 1
  New or worsened to grade 4 (Parameter: blood bilirubin increased): number analyzed (Participants) | 154 | 40
  New or worsened to grade 4 (Parameter: blood bilirubin increased) | 0 | 0
  New or worsened to grade 1 (Parameter: creatine phosphokinase [CPK] increased): number analyzed (Participants) | 151 | 41
  New or worsened to grade 1 (Parameter: creatine phosphokinase [CPK] increased) | 22 | 3
  New or worsened to grade 2 (Parameter: CPK increased): number analyzed (Participants) | 151 | 41
  New or worsened to grade 2 (Parameter: CPK increased) | 8 | 1
  New or worsened to grade 3 (Parameter: CPK increased): number analyzed (Participants) | 151 | 41
  New or worsened to grade 3 (Parameter: CPK increased) | 2 | 3
  New or worsened to grade 4 (Parameter: CPK increased): number analyzed (Participants) | 151 | 41
  New or worsened to grade 4 (Parameter: CPK increased) | 0 | 1
  New or worsened to grade 1 (Parameter: creatinine increased): number analyzed (Participants) | 153 | 40
  New or worsened to grade 1 (Parameter: creatinine increased) | 87 | 24
  New or worsened to grade 2 (Parameter: creatinine increased): number analyzed (Participants) | 153 | 40
  New or worsened to grade 2 (Parameter: creatinine increased) | 12 | 4
  New or worsened to grade 3 (Parameter: creatinine increased): number analyzed (Participants) | 153 | 40
  New or worsened to grade 3 (Parameter: creatinine increased) | 1 | 0
  New or worsened to grade 4 (Parameter: creatinine increased): number analyzed (Participants) | 153 | 40
  New or worsened to grade 4 (Parameter: creatinine increased) | 1 | 0
  New or worsened to grade 1 (Parameter: gamma glutamyl transferase [GGT] increased): number analyzed (Participants) | 147 | 40
  New or worsened to grade 1 (Parameter: gamma glutamyl transferase [GGT] increased) | 23 | 8
  New or worsened to grade 2 (Parameter: GGT increased): number analyzed (Participants) | 147 | 40
  New or worsened to grade 2 (Parameter: GGT increased) | 16 | 5
  New or worsened to grade 3 (Parameter: GGT increased): number analyzed (Participants) | 147 | 40
  New or worsened to grade 3 (Parameter: GGT increased) | 26 | 7
  New or worsened to grade 4 (Parameter: GGT increased): number analyzed (Participants) | 147 | 40
  New or worsened to grade 4 (Parameter: GGT increased) | 1 | 1
  New or worsened to grade 1 (Parameter: hypercalcemia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 1 (Parameter: hypercalcemia) | 11 | 4
  New or worsened to grade 2 (Parameter: hypercalcemia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 2 (Parameter: hypercalcemia) | 0 | 0
  New or worsened to grade 3 (Parameter: hypercalcemia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 3 (Parameter: hypercalcemia) | 1 | 0
  New or worsened to grade 4 (Parameter: hypercalcemia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 4 (Parameter: hypercalcemia) | 0 | 0
  New or worsened to grade 1 (Parameter: hyperglycemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 1 (Parameter: hyperglycemia) | 23 | 5
  New or worsened to grade 2 (Parameter: hyperglycemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 2 (Parameter: hyperglycemia) | 2 | 0
  New or worsened to grade 3 (Parameter: hyperglycemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 3 (Parameter: hyperglycemia) | 3 | 2
  New or worsened to grade 4 (Parameter: hyperglycemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 4 (Parameter: hyperglycemia) | 1 | 0
  New or worsened to grade 1 (Parameter: hyperkalemia): number analyzed (Participants) | 156 | 40
  New or worsened to grade 1 (Parameter: hyperkalemia) | 13 | 3
  New or worsened to grade 2 (Parameter: hyperkalemia): number analyzed (Participants) | 156 | 40
  New or worsened to grade 2 (Parameter: hyperkalemia) | 6 | 0
  New or worsened to grade 3 (Parameter: hyperkalemia): number analyzed (Participants) | 156 | 40
  New or worsened to grade 3 (Parameter: hyperkalemia) | 1 | 0
  New or worsened to grade 4 (Parameter: hyperkalemia): number analyzed (Participants) | 156 | 40
  New or worsened to grade 4 (Parameter: hyperkalemia) | 1 | 0
  New or worsened to grade 1 (Parameter: hypermagnesemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 1 (Parameter: hypermagnesemia) | 9 | 4
  New or worsened to grade 2 (Parameter: hypermagnesemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 2 (Parameter: hypermagnesemia) | 0 | 0
  New or worsened to grade 3 (Parameter: hypermagnesemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 3 (Parameter: hypermagnesemia) | 3 | 0
  New or worsened to grade 4 (Parameter: hypermagnesemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 4 (Parameter: hypermagnesemia) | 0 | 0
  New or worsened to grade 1 (Parameter: hypernatremia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 1 (Parameter: hypernatremia) | 8 | 1
  New or worsened to grade 2 (Parameter: hypernatremia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 2 (Parameter: hypernatremia) | 0 | 0
  New or worsened to grade 3 (Parameter: hypernatremia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 3 (Parameter: hypernatremia) | 0 | 0
  New or worsened to grade 4 (Parameter: hypernatremia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 4 (Parameter: hypernatremia) | 0 | 0
  New or worsened to grade 1 (Parameter: hypoalbuminemia): number analyzed (Participants) | 150 | 39
  New or worsened to grade 1 (Parameter: hypoalbuminemia) | 21 | 6
  New or worsened to grade 2 (Parameter: hypoalbuminemia): number analyzed (Participants) | 150 | 39
  New or worsened to grade 2 (Parameter: hypoalbuminemia) | 10 | 2
  New or worsened to grade 3 (Parameter: hypoalbuminemia): number analyzed (Participants) | 150 | 39
  New or worsened to grade 3 (Parameter: hypoalbuminemia) | 2 | 1
  New or worsened to grade 4 (Parameter: hypoalbuminemia): number analyzed (Participants) | 150 | 39
  New or worsened to grade 4 (Parameter: hypoalbuminemia) | 0 | 0
  New or worsened to grade 1 (Parameter: hypocalcemia): number analyzed (Participants) | 153 | 41
  New or worsened to grade 1 (Parameter: hypocalcemia) | 27 | 2
  New or worsened to grade 2 (Parameter: hypocalcemia): number analyzed (Participants) | 153 | 41
  New or worsened to grade 2 (Parameter: hypocalcemia) | 6 | 1
  New or worsened to grade 3 (Parameter: hypocalcemia): number analyzed (Participants) | 153 | 41
  New or worsened to grade 3 (Parameter: hypocalcemia) | 3 | 0
  New or worsened to grade 4 (Parameter: hypocalcemia): number analyzed (Participants) | 153 | 41
  New or worsened to grade 4 (Parameter: hypocalcemia) | 0 | 0
  New or worsened to grade 1 (Parameter: hypoglycemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 1 (Parameter: hypoglycemia) | 10 | 4
  New or worsened to grade 2 (Parameter: hypoglycemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 2 (Parameter: hypoglycemia) | 1 | 0
  New or worsened to grade 3 (Parameter: hypoglycemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 3 (Parameter: hypoglycemia) | 0 | 0
  New or worsened to grade 4 (Parameter: hypoglycemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 4 (Parameter: hypoglycemia) | 0 | 0
  New or worsened to grade 1 (Parameter: hypokalemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 1 (Parameter: hypokalemia) | 0 | 0
  New or worsened to grade 2 (Parameter: hypokalemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 2 (Parameter: hypokalemia) | 24 | 8
  New or worsened to grade 3 (Parameter: hypokalemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 3 (Parameter: hypokalemia) | 4 | 1
  New or worsened to grade 4 (Parameter: hypokalemia): number analyzed (Participants) | 155 | 41
  New or worsened to grade 4 (Parameter: hypokalemia) | 0 | 0
  New or worsened to grade 1 (Parameter: hypomagnesemia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 1 (Parameter: hypomagnesemia) | 24 | 5
  New or worsened to grade 2 (Parameter: hypomagnesemia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 2 (Parameter: hypomagnesemia) | 2 | 0
  New or worsened to grade 3 (Parameter: hypomagnesemia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 3 (Parameter: hypomagnesemia) | 1 | 0
  New or worsened to grade 4 (Parameter: hypomagnesemia): number analyzed (Participants) | 156 | 41
  New or worsened to grade 4 (Parameter: hypomagnesemia) | 1 | 0
  New or worsened to grade 1 (Parameter: hyponatremia): number analyzed (Participants) | 153 | 40
  New or worsened to grade 1 (Parameter: hyponatremia) | 29 | 10
  New or worsened to grade 2 (Parameter: hyponatremia): number analyzed (Participants) | 153 | 40
  New or worsened to grade 2 (Parameter: hyponatremia) | 0 | 0
  New or worsened to grade 3 (Parameter: hyponatremia): number analyzed (Participants) | 153 | 40
  New or worsened to grade 3 (Parameter: hyponatremia) | 11 | 2
  New or worsened to grade 4 (Parameter: hyponatremia): number analyzed (Participants) | 153 | 40
  New or worsened to grade 4 (Parameter: hyponatremia) | 0 | 0
  New or worsened to grade 1 (Parameter: hypophosphatemia): number analyzed (Participants) | 153 | 41
  New or worsened to grade 1 (Parameter: hypophosphatemia) | 0 | 0
  New or worsened to grade 2 (Parameter: hypophosphatemia): number analyzed (Participants) | 153 | 41
  New or worsened to grade 2 (Parameter: hypophosphatemia) | 18 | 4
  New or worsened to grade 3 (Parameter: hypophosphatemia): number analyzed (Participants) | 153 | 41
  New or worsened to grade 3 (Parameter: hypophosphatemia) | 2 | 1
  New or worsened to grade 4 (Parameter: hypophosphatemia): number analyzed (Participants) | 153 | 41
  New or worsened to grade 4 (Parameter: hypophosphatemia) | 0 | 0
  New or worsened to grade 1 (Parameter: lipase increased): number analyzed (Participants) | 157 | 41
  New or worsened to grade 1 (Parameter: lipase increased) | 13 | 4
  New or worsened to grade 2 (Parameter: lipase increased): number analyzed (Participants) | 157 | 41
  New or worsened to grade 2 (Parameter: lipase increased) | 9 | 3
  New or worsened to grade 3 (Parameter: lipase increased): number analyzed (Participants) | 157 | 41
  New or worsened to grade 3 (Parameter: lipase increased) | 7 | 2
  New or worsened to grade 4 (Parameter: lipase increased): number analyzed (Participants) | 157 | 41
  New or worsened to grade 4 (Parameter: lipase increased) | 2 | 1
  New or worsened to grade 1 (Parameter: serum amylase increased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 1 (Parameter: serum amylase increased) | 16 | 3
  New or worsened to grade 2 (Parameter: serum amylase increased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 2 (Parameter: serum amylase increased) | 1 | 2
  New or worsened to grade 3 (Parameter: serum amylase increased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 3 (Parameter: serum amylase increased) | 2 | 2
  New or worsened to grade 4 (Parameter: serum amylase increased): number analyzed (Participants) | 156 | 41
  New or worsened to grade 4 (Parameter: serum amylase increased) | 1 | 1

5. Secondary Outcome: Serum Lowest (Trough) Concentration (Ctrough) of Avelumab
Description: Ctrough was defined as predose concentration during multiple dosing. The determination method of Ctrough was observing directly from data. The lower limit of quantification (LLQ) was 0.2 mcg/mL. For Cycle 1 Day 1, as the number of observations above lower limit of quantification (NALQ) = 0, summary statistics were not presented.
Time Frame: Predose on Day 1 of Cycles 1, 3, 6, 12, 18, 24 and Day 15 of Cycle 1
Population: The avelumab PK concentration analysis set included all participants (Cohort 1 and Cohort 2 combined) who received at least 1 dose of study intervention and had at least one concentration measurement for avelumab. Number of participants analyzed = number of participants evaluable for this OM. Number analyzed = participants evaluable at the specific time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram(mcg)/milliliter(mL)
Groups:
- Avelumab 800 mg Intravenous (IV) Q2W Plus Talazoparib: Talazoparib was self-administered orally at a starting dose of 1 mg QD for participants with normal renal function or mild renal impairment until End of Treatment. Participants with moderate renal impairment received starting dose of 0.75 mg QD. Avelumab was administered as a 1-hour IV infusion Q2W on Days 1 and 15 of each 28-day cycle at a dose of 800 mg after administration of talazoparib and the premedication.
Arm/Group | Avelumab 800 mg Intravenous (IV) Q2W Plus Talazoparib
Number analyzed (Participants) | 199
microgram(mcg)/milliliter(mL)
  CYCLE1DAY1: number analyzed (Participants) | 180
  CYCLE1DAY1 | NA (NA) — Summary statistics were not presented for NALQ = 0.
  CYCLE1DAY15: number analyzed (Participants) | 164
  CYCLE1DAY15 | 21.06 (58)
  CYCLE3DAY1: number analyzed (Participants) | 110
  CYCLE3DAY1 | 32.65 (63)
  CYCLE6DAY1: number analyzed (Participants) | 83
  CYCLE6DAY1 | 36.23 (60)
  CYCLE12DAY1: number analyzed (Participants) | 35
  CYCLE12DAY1 | 41.80 (60)
  CYCLE18DAY1: number analyzed (Participants) | 16
  CYCLE18DAY1 | 35.19 (54)
  CYCLE24DAY1: number analyzed (Participants) | 10
  CYCLE24DAY1 | 37.21 (54)

6. Secondary Outcome: Serum Maximum Concentration (Cmax) for Avelumab
Description: Cmax was defined as maximum observed plasma concentration. The determination method of Cmax was observing directly from data.
Time Frame: One hour post-dose on Day 1 of Cycles 1, 3, 6, 12, 18, 24 and Day 15 of Cycle 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Groups:
- Avelumab 800 mg IV Q2W Plus Talazoparib: Talazoparib was self-administered orally at a starting dose of 1 mg QD for participants with normal renal function or mild renal impairment until End of Treatment. Participants with moderate renal impairment received starting dose of 0.75 mg QD. Avelumab was administered as a 1-hour IV infusion Q2W on Days 1 and 15 of each 28-day cycle at a dose of 800 mg after administration of talazoparib and the premedication.
Arm/Group | Avelumab 800 mg IV Q2W Plus Talazoparib
Number analyzed (Participants) | 199
mcg/mL
  CYCLE1DAY1: number analyzed (Participants) | 161
  CYCLE1DAY1 | 223.0 (39)
  CYCLE1DAY15: number analyzed (Participants) | 146
  CYCLE1DAY15 | 221.6 (38)
  CYCLE3DAY1: number analyzed (Participants) | 114
  CYCLE3DAY1 | 225.6 (34)
  CYCLE6DAY1: number analyzed (Participants) | 79
  CYCLE6DAY1 | 222.3 (37)
  CYCLE12DAY1: number analyzed (Participants) | 35
  CYCLE12DAY1 | 248.2 (25)
  CYCLE18DAY1: number analyzed (Participants) | 17
  CYCLE18DAY1 | 265.9 (20)
  CYCLE24DAY1: number analyzed (Participants) | 9
  CYCLE24DAY1 | 286.1 (21)

7. Secondary Outcome: Plasma Ctrough for Talazoparib
Description: Ctrough was defined as predose concentration during multiple dosing. The determination method of Ctrough was observing directly from data. The lower limit of quantification (LLQ) was 25 pg/mL. For Cycle 1 Day 1, as the number of observations above lower limit of quantification (NALQ) = 0, summary statistics were not presented. Evaluable participants were participants with non-missing Ctrough concentrations at each specific time point and meeting 2 conditions: participants received 14 consecutive days of talazoparib dose without dosing interruption prior to sample collection (except on Cycle 1 Day 1) and sample collection within 24 hours ± 10% (2 hours and 24 minutes) after the previous day's dose and no more than 5 minutes (0.083 hours) after the administration of the dose on the day of PK sample collection. Predose PK samples on Cycle 1 Day 1 must have been collected prior to dose.
Time Frame: Predose on Cycle 1 Days 1, 15 and Cycle 3 Day 1
Population: The talazoparib PK concentration analysis set included all participants (Cohort 1 and Cohort 2 combined) who received at least 1 dose of study intervention and had at least one Ctrough concentration measurement for talazoparib. Number of participants analyzed = number of participants evaluable for this OM. Number analyzed = participants evaluable at the specific time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram(pg)/mL
Arm/Group | Avelumab 800 mg IV Q2W Plus Talazoparib
Number analyzed (Participants) | 199
picogram(pg)/mL
  CYCLE1DAY1 (Starting Dose: 1 mg QD): number analyzed (Participants) | 170
  CYCLE1DAY1 (Starting Dose: 1 mg QD) | NA (NA) — Summary statistics were not presented for NALQ = 0.
  CYCLE1DAY15 (Starting Dose: 1 mg QD): number analyzed (Participants) | 62
  CYCLE1DAY15 (Starting Dose: 1 mg QD) | 4649 (61)
  CYCLE3DAY1 (Starting Dose: 1 mg QD): number analyzed (Participants) | 30
  CYCLE3DAY1 (Starting Dose: 1 mg QD) | 3313 (113)
  CYCLE1DAY1 (Starting Dose: 0.75 mg QD): number analyzed (Participants) | 16
  CYCLE1DAY1 (Starting Dose: 0.75 mg QD) | NA (NA) — Summary statistics were not presented for NALQ = 0.
  CYCLE1DAY15 (Starting Dose: 0.75 mg QD): number analyzed (Participants) | 2
  CYCLE1DAY15 (Starting Dose: 0.75 mg QD) | 7612 (NA) — Geometric Coefficient of Variation was not estimable due to insufficient number of participants with results.
  CYCLE3DAY1 (Starting Dose: 0.75 mg QD): number analyzed (Participants) | 4
  CYCLE3DAY1 (Starting Dose: 0.75 mg QD) | 4314 (42)

8. Secondary Outcome: Plasma Post-dose Concentrations for Talazoparib
Description: In this OM, the post-dose concentrations for talazoparib in plasma were reported.
Time Frame: Postdose (samples collected within 2 hours post dose plus/minus 12 minutes) on Days 1,15 of Cycle 1, and Day 1 of Cycle 3
Population: The Analysis Population included all participants (Cohort 1 and Cohort 2 combined) who received at least 1 dose of talazoparib, had at least one non-missing concentration measurement at any collection scheduled time point, received 14 consecutive days of talazoparib dose without dosing interruption prior to sample collection (except on Cycle 1 Day 1) and sample collection was performed within ± 10% (12 minutes) of nominal time post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Avelumab 800 mg IV Q2W Plus Talazoparib
Number analyzed (Participants) | 106
pg/mL
  CYCLE1DAY1 (Starting Dose: 1 mg QD): number analyzed (Participants) | 76
  CYCLE1DAY1 (Starting Dose: 1 mg QD) | 1833 (275)
  CYCLE1DAY15 (Starting Dose: 1 mg QD): number analyzed (Participants) | 51
  CYCLE1DAY15 (Starting Dose: 1 mg QD) | 7985 (79)
  CYCLE3DAY1 (Starting Dose: 1 mg QD): number analyzed (Participants) | 22
  CYCLE3DAY1 (Starting Dose: 1 mg QD) | 7800 (69)
  CYCLE1DAY1 (Starting Dose: 0.75 mg QD): number analyzed (Participants) | 6
  CYCLE1DAY1 (Starting Dose: 0.75 mg QD) | 1663 (100)
  CYCLE1DAY15 (Starting Dose: 0.75 mg QD): number analyzed (Participants) | 6
  CYCLE1DAY15 (Starting Dose: 0.75 mg QD) | 12590 (47)
  CYCLE3DAY1 (Starting Dose: 0.75 mg QD): number analyzed (Participants) | 3
  CYCLE3DAY1 (Starting Dose: 0.75 mg QD) | 8366 (53)

9. Secondary Outcome: Number of Participants by Avelumab Anti-drug Antibody (ADA) Categories
Description: Blood samples were assayed for ADA using a validated assay. ADA never-positive = no positive ADA results at any time point. ADA ever-positive =at least one positive ADA result at any time point. Baseline ADA positive =a positive ADA result at baseline. Treatment-boosted ADA =a positive ADA result at baseline and the titer >=8×baseline titer at least once after treatment with avelumab. Treatment-induced ADA = participant was ADA-negative at baseline and had at least one positive post-baseline ADA result; or the participant had at least one positive post-baseline ADA result if no baseline sample. Transient ADA response = participants with treatment-induced ADA had (a single positive ADA result or duration between first and last positive result <16 weeks) and ADA result at the last assessment was not positive. Persistent ADA response =participants with treatment-induced ADA had duration between first and last positive ADA result >=16 weeks or a positive ADA result at the last assessment.
Time Frame: Predose (within 2 hours before start of avelumab infusion) on Day 1 of Cycles 1, 3, 6, 12, 18, 24 and Day 15 of Cycle 1
Population: Number of Participants Analyzed = participants in the immunogenicity analysis set who had at least 1 ADA sample collected for avelumab. Number Analyzed (N0) = participants with at least one valid ADA result at any time point; (N1) = participants with valid baseline ADA result; (N2) = participants with valid baseline ADA results and at least one valid post-baseline ADA result; (N3) = participants with at least one valid post-baseline ADA result and without positive baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 40
Participants
  ADA never-positive (n/N0) | 153 | 39
  ADA ever-positive (n/N0) | 6 | 1
  Baseline ADA positive (n/N1): number analyzed (Participants) | 150 | 38
  Baseline ADA positive (n/N1) | 5 | 1
  Treatment-boosted ADA (n/N2): number analyzed (Participants) | 143 | 37
  Treatment-boosted ADA (n/N2) | 0 | 0
  Treatment-induced ADA (n/N3): number analyzed (Participants) | 147 | 38
  Treatment-induced ADA (n/N3) | 1 | 0
  Transient ADA response (n/N3): number analyzed (Participants) | 147 | 38
  Transient ADA response (n/N3) | 1 | 0
  Persistent ADA response (n/N3): number analyzed (Participants) | 147 | 38
  Persistent ADA response (n/N3) | 0 | 0

10. Secondary Outcome: Number of Participants With Neutralizing Antibodies (Nab) Levels Against Avelumab Ever-Positive
Description: Nab ever-positive was defined as at least one positive Nab result at any time point. Samples positive for ADA with persistent treatment-induced ADA response could be analyzed for Nab.
Time Frame: Predose (within 2 hours before start of avelumab infusion) on Day 1 of Cycles 1, 3, 6, 12, 18, 24 and Day 15 of Cycle 1
Population: The immunogenicity analysis set included participants who had at least 1 Nab sample collected for avelumab. Nabs data were not collected due to insufficient number of participants with persistent treatment-induced ADA response. Therefore, the number of participants analyzed for this OM was 0.
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage of Participants With Confirmed OR as Assessed by The Investigator
Description: For participants with solid tumors, except mCRPC, OR was defined as a CR or PR per RECIST v1.1, both confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. For participants with mCRPC, OR was defined as the percentage of participants with a best overall soft tissue response of CR or PR per RECIST v1.1 with no evidence of confirmed bone disease progression per PCWG3 criteria. Per RECIST v1.1, CR was defined as complete disappearance of all target and non-target lesions with the exception of nodal disease. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. Non-target PR lesions must be non-PD, where PD was unequivocal progression of pre-existing lesions.
Time Frame: From the first dose of study treatment until the date of first documented disease progression or date of death from any cause, whichever comes first, assessed up to approximately 24 months
Population: All efficacy analyses were performed based on the full analysis set. The full analysis set included all enrolled participants who received at least 1 dose of study treatment. Participants were classified according to the cohort assigned at enrollment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Percentage of participants | 34.6 [27.2 to 42.5] | 14.6 [5.6 to 29.2]

12. Secondary Outcome: Time to Tumor Response (TTR) as Assessed by BICR
Description: For participants with solid tumors, except mCRPC: TTR was defined for participants with confirmed objective response (CR or PR) as the time from the first dose of study treatment to the first documentation of objective tumor response. For participants with mCRPC: TTR was defined as the time from the first dose of study treatment to the first objective evidence of soft tissue response with no evidence of confirmed bone disease progression on bone scan per PCWG3. Soft tissue response was defined as a Best Overall Response (BOR) of CR or PR per RECIST v1.1.
Time Frame: Baseline up to approximately 24 months
Population: The analysis population included all enrolled participants who received at least 1 dose of study treatment and with confirmed CR or PR as assessed by BICR.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 44 | 3
Months | 1.82 [1.5 to 12.1] | 5.52 [1.6 to 16.8]

13. Secondary Outcome: TTR as Assessed by Investigator
Description: For participants with solid tumors, except mCRPC: TTR was defined for participants with confirmed objective response (CR or PR) as the time from the first dose of study treatment to the first documentation of objective tumor response. For participants with mCRPC: TTR was defined as the time from the first dose of study treatment to the first objective evidence of soft tissue response with no evidence of confirmed bone disease progression on bone scan per PCWG3. Soft tissue response was defined as a BOR of CR or PR per RECIST v1.1.
Time Frame: Baseline up to approximately 24 months
Population: The analysis population included all enrolled participants who received at least 1 dose of study treatment and with confirmed CR or PR as assessed by investigator.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 55 | 6
Months | 1.84 [1.5 to 18.4] | 3.99 [1.9 to 14.0]

14. Secondary Outcome: Duration of Response (DoR) as Assessed by BICR
Description: For participants with solid tumors, except mCRPC: DoR was defined for participants with confirmed objective response (CR or PR) as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occured first. For participants with mCRPC: DoR was defined for participants with confirmed objective response (CR or PR) as the time from the first objective evidence of soft tissue response (subsequently confirmed) per RECIST v1.1 and no evidence of confirmed bone disease progression by PCWG3 to the first subsequent objective evidence of radiographic progression or death due to any cause, whichever occured first. Radiographic progression was defined as soft tissue progression evaluated per RECIST v1.1 or bone disease progression evaluated per PCWG3.
Time Frame: Baseline up to approximately 24 months
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 44 | 3
Months | 12.5 [7.5 to NA] — The reason for NA is that the upper limit of the confidence interval is not crossing the 50% bound. | NA [6.7 to NA] — The reason for NA is that the median and upper limit of the confidence interval are not crossing the 50% bound.

15. Secondary Outcome: DoR as Assessed by Investigator
Description: For participants with solid tumors, except mCRPC: DoR was defined for participants with confirmed objective response (CR or PR) as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. For participants with mCRPC: DoR was defined for participants with confirmed objective response (CR or PR) as the time from the first objective evidence of soft tissue response (subsequently confirmed) per RECIST v1.1 and no evidence of confirmed bone disease progression by PCWG3 to the first subsequent objective evidence of radiographic progression or death due to any cause, whichever occurred first. Radiographic progression was defined as soft tissue progression evaluated per RECIST v1.1 or bone disease progression evaluated per PCWG3.
Time Frame: Baseline up to approximately 24 months
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 55 | 6
Months | 8.8 [7.5 to 10.7] | 7.1 [5.5 to 9.7]

16. Secondary Outcome: Progression Free Survival (PFS) as Assessed by BICR
Description: For participants with solid tumors, except mCRPC: PFS was defined as the time from the first dose of study treatment to the date of disease progression by RECIST v1.1 or death due to any cause, whichever occurred first. For participants with mCRPC: PFS was defined as the time from the first dose of study treatment to documentation of radiographic progression in soft tissue evaluated per RECIST v1.1, in bone evaluated per PCWG3, or death, whichever occurred first.
Time Frame: Baseline up to approximately 24 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Months | 3.7 [3.1 to 5.4] | 3.5 [1.8 to 5.5]

17. Secondary Outcome: PFS as Assessed by Investigator
Description: as for outcome 16
Time Frame: Baseline up to approximately 24 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Months | 5.3 [3.7 to 5.6] | 3.7 [2.1 to 7.4]

18. Secondary Outcome: Overall Survival (OS) for All Participants
Description: OS was defined as the time from the first dose of study treatment to the date of death. Participants without an event (death) were censored at the date of last contact.
Time Frame: Baseline up to approximately 24 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Months | 11.9 [10.1 to 13.7] | 16.4 [12.8 to 21.9]

19. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression for Participants With mCRPC
Description: For participants with mCRPC, time to PSA progression was defined as the time from the first dose to the date that a >=25% increase in PSA with an absolute increase of >=2 μg/L (2 ng/mL) above the nadir (or baseline for participants with no PSA decline) was documented, confirmed by a second consecutive PSA value obtained >=3 weeks (21 days) later.
Time Frame: Baseline up to approximately 24 months
Population: The analysis population included all participants with mCRPC who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 26 | 5
Months | 6.5 [3.7 to 12.7] | 11.3 [3.7 to NA] — The upper limit of the confidence interval is not crossing the 50% bound.

20. Secondary Outcome: Number of Participants With Confirmed PSA Response
Description: For participants with mCRPC, PSA response was defined as confirmed PSA decline >=50% compared to baseline. PSA response was calculated as a decline from baseline PSA (ng/mL) to the maximal PSA response with a threshold of 50%. A PSA response must have been confirmed by a second consecutive value at least 3 weeks later.
Time Frame: Baseline up to approximately 24 months
Population: The analysis population included all participants with mCRPC who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 26 | 5
Participants | 17 | 2

21. Secondary Outcome: Number of Participants With Circulating Tumor Cell (CTC) Count Conversion
Description: For participants with mCRPC, CTC count conversion was defined as a decrease in CTC count from >=5 CTC per 7.5 mL of blood at baseline to <5 CTC per 7.5 mL of blood anytime on study.
Time Frame: Day 1 of Cycle 1 to Cycle 4
Population: The analysis population included all enrolled participants with mCRPC who received at least 1 dose of study treatment, and with CTC count >=5 CTC per 7.5 mL of blood at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 13 | 2
Participants | 11 | 1

22. Secondary Outcome: Number of Participants With Cancer Antigen 125 (CA-125) Response
Description: For participants with ovarian cancer, CA-125 response was defined as at least a 50% reduction in CA-125 levels from baseline. The response must have been confirmed and maintained for at least 28 days.
Time Frame: Baseline, Day 1 of each treatment Cycle, maximum up to 4.3 years approximately
Population: The analysis population included all participants with ovarian cancer who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 26 | 3
Participants | 9 | 0

23. Secondary Outcome: Number of Participants With Positive Programmed Death Ligand 1 (PD-L1) Expression in Baseline Tumor Tissue
Description: PD-L1 expression on tumor and infiltrating immune cells was measured by immunohistochemistry (IHC). PD-L1 expression level was defined as the number of PD-L1 positive cells and/or qualitative assessment of PD-L1 staining on tumor and inflammatory cells in regions of interest. This OM reported the number of participants classified as positive according to scoring algorithms and cut-offs established from external sources.
Time Frame: Baseline
Population: The biomarker analysis set included all participants who received at least 1 dose of study treatment and had at least 1 screening biomarker assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Participants | 27 | 0

24. Secondary Outcome: Number of Participants With Different Status for Defects in BRCA1, BRCA2 and ATM
Description: Participants were enrolled in the two cohorts based on BRCA 1/2 and ATM defect status assessed by the local laboratory. The participant BRCA and ATM status was assessed retrospectively by central laboratory, that may differ from the status assessed by the local laboratory. The ATM participants with a negative ATM status per the central laboratory were reported to have a positive ATM status per the local laboratory. Therefore, participants with negative ATM status might have been included in the ATM defect cohort. For defects in BRCA1, BRCA2 and ATM by central laboratory analysis, participants were classified as positive, negative, not analyzable or missing. The number of participants in each category of BRCA 1 defect, BRCA 2 defect, BRCA 1 or BRCA 2 defect and ATM defect were presented.
Time Frame: Baseline
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Participants
  BRCA1 status: Positive | 52 | 0
  BRCA1 status: Negative | 65 | 29
  BRCA1 status: Not analyzable | 21 | 4
  BRCA1 status: Missing | 21 | 8
  BRCA2 status: Positive | 53 | 1
  BRCA2 status: Negative | 64 | 28
  BRCA2 status: Not analyzable | 21 | 4
  BRCA2 status: Missing | 21 | 8
  BRCA status: Positive | 105 | 1
  BRCA status: Negative | 12 | 28
  BRCA status: Not analyzable | 21 | 4
  BRCA status: Missing | 21 | 8
  ATM status: Positive | 2 | 26
  ATM status: Negative | 115 | 3
  ATM status: Not analyzable | 21 | 4
  ATM status: Missing | 21 | 8

25. Secondary Outcome: Number of Participants by Status of Tumor Mutational Burden (TMB) at Baseline
Description: TMB was defined as the total number of mutations in the tumor genome, or number of mutations per megabase of DNA if derived from targeted sequencing. TMB categories were defined as high, low for a number of mutations per megabase >=10 and <10, respectively. The TMB category 'Not analyzable' included participants with available samples but not evaluable. The TMB category 'Missing' included participants with no sample available. The number of participants in each category at only baseline were tabulated.
Time Frame: Baseline
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
Number analyzed (Participants) | 159 | 41
Participants
  TMB status high | 9 | 2
  TMB status low | 95 | 23
  TMB status not analyzable | 34 | 8
  TMB status missing | 21 | 8

ADVERSE EVENTS:
Time Frame: From baseline up to 30 days after last dose of study treatment, maximum up to 4.3 years approximately.
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Cohort 1 (BRCA 1/2 Defect) | Cohort 2 (ATM Defect)
All-Cause Mortality (participants affected / at risk) | 15/159 | 3/41
Serious Adverse Events (participants affected / at risk) | 50/159 | 7/41
Other Adverse Events (participants affected / at risk) | 153/159 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (BRCA 1/2 Defect) (N=159) | Cohort 2 (ATM Defect) (N=41)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Bone marrow disorder (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Small intestine polyp (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Disease progression (General disorders) | 8 | 2
Pyrexia (General disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Bacterial abdominal infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 1
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (BRCA 1/2 Defect) (N=159) | Cohort 2 (ATM Defect) (N=41)
Anaemia (Blood and lymphatic system disorders) | 81 | 18
Neutropenia (Blood and lymphatic system disorders) | 20 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 5
Hypothyroidism (Endocrine disorders) | 10 | 5
Abdominal distension (Gastrointestinal disorders) | 5 | 6
Abdominal pain (Gastrointestinal disorders) | 30 | 6
Ascites (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 39 | 8
Diarrhoea (Gastrointestinal disorders) | 36 | 10
Dyspepsia (Gastrointestinal disorders) | 10 | 3
Nausea (Gastrointestinal disorders) | 73 | 21
Vomiting (Gastrointestinal disorders) | 39 | 11
Asthenia (General disorders) | 27 | 2
Chills (General disorders) | 17 | 5
Fatigue (General disorders) | 50 | 19
Influenza like illness (General disorders) | 10 | 2
Oedema peripheral (General disorders) | 12 | 4
Pyrexia (General disorders) | 28 | 3
Sinusitis (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 12 | 3
Urinary tract infection (Infections and infestations) | 11 | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 22 | 3
Alanine aminotransferase increased (Investigations) | 16 | 7
Aspartate aminotransferase increased (Investigations) | 18 | 6
Blood bilirubin increased (Investigations) | 8 | 3
Blood creatine phosphokinase increased (Investigations) | 7 | 4
Blood creatinine increased (Investigations) | 3 | 5
Gamma-glutamyltransferase increased (Investigations) | 9 | 3
Lymphocyte count decreased (Investigations) | 2 | 3
Neutrophil count decreased (Investigations) | 21 | 5
Platelet count decreased (Investigations) | 25 | 11
Weight decreased (Investigations) | 10 | 2
White blood cell count decreased (Investigations) | 12 | 4
Decreased appetite (Metabolism and nutrition disorders) | 33 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Dizziness (Nervous system disorders) | 19 | 1
Headache (Nervous system disorders) | 35 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 21 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 1
Hot flush (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT03565991/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03565991/SAP_001.pdf